CLINICAL TRIAL: NCT01706757
Title: Assessment of Motivity in People Aged 65 to 86 Years : Comparison of a Standard Assessment Versus a Technological Solution
Brief Title: Assessment of Motivity in People Aged 65 to 86 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Clinical Research and Innovation (Other)
Responsible Party: Sponsor-Investigator, Department of Clinical Research and Innovation, Department of Clinical Research and Innovation (drc), Centre Hospitalier Universitaire de Nice
Organization: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 11-PP-05
Record Dates: First submitted 2012-06-18; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-07

CONDITIONS: Assessment of Motivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with go-cart (Experimental): conducts exercises with the help of a go-cart
  Interventions: Device: go-cart
- without go-cart (No Intervention): conduct exercises without go-cart

INTERVENTIONS:
Device: go-cart — conducts exercises with the help of a go-cart
  Arms: with go-cart

SUMMARY:
The ability to walk is one of the fundamental attributes of human beings. However, with advancing age this ability is modified by a combination of physiological and pathological aging.These changes mainly involve an irregularity of the pitch, reducing the length of the stride, instability and a decrease in walking speed (Beauchet et al., 2002). Tinetti, Speecheley, Ginter (1988, from Ch Wider, F. Vingerhoets, J Bogousslavsky, 2005) show that 20-30% of heathly older fall each year and state that one of these falls, 25% result in injuries with significant effect and 5% a fracture. In addition to the risk of fracture fear of falling exists in many older people even before a drop in effective (Recommandation of HAS, 2005).In France, about 9 000 deaths of people aged over 65 are associated each year with a fall and this association increases rapidly with advancing age in both sexes. It is therefore important in terms of public health, learn to recognize the gait disturbance, to prevent and to make adequate assessments to reduce the risk of falls. Tools exist to assess the risk of falling. Some are comprehensive but time-consuming and are generally discarded in favour of other simpler tests (test of Tinetti or get up and go test). However, the listing of these lacks precision, particularly in terms of duration single timer.To overcome these biases, innovative technology solutions seem to be a good way. In this study, the investigators will use the motorized go-cart developed by INRIA, entitled ANG (for Assisted Navigation Guide), to obtain more reliable and accurate measurements of parameters such as walking speed and direction. Thus, the investigators set the main objective, to compare a standard evaluation of the process to a technology assessment, in participants aged 65 to 86 years. And as secondary objectives : evaluate the acceptance of using go-cart ANG in the elderly, develop an index of walking and test the feasibility of detecting a weakness of the knee joint by ANG undetected at clinic.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged between 65 and 86 years
* participants with no locomotor disability hindering the implementation of the protocol
* participants with no global cognitive impairment (MMSE score <24) (Folstein et al. 1975), or arguments in favor of the following diagnoses : probable Alzheimer's disease according to the criteria of the NINCDS-ADRDA, major depressive episode according to DSM-IV-R
* participant with no apathy according to diagnostic criteria for apathy (Robert, Onyike et al. 2009)
* participants recipients of social security
* signature of informed consent.

Exclusion Criteria:

* impossibility of carrying out the experimental protocol because of a mobility impairment

Ages: 65 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Walking speed. | one day
  Walking speed. This will be calculated from an exercise where participants will be asked to walk from one point to another of the room according to the instructions set out below.
  The average speed of walking in technology assessment, will be directly collected by ANG.
  A comparison of estimated speeds as standard and technology can then be performed.

SECONDARY OUTCOMES:
acceptance of the go-cart | one day
  1. to assess the acceptance of ANG in the elderly. A questionnaire after the experiment will determine the level of acceptance of the go-cart, and to assess its ease of use.
  2. Develop mathematical algorithms to index certain characteristics of the market depending on the linear trajectory, U-turns. c) The detection of a weak joint. d) The index of walking on a path set will be made with and without use of the go-cart. e) Evaluate the ability of subjects to perform complex and precise trajectories

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Robert, Md, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Centre Mémoire de Ressources et de Recherche, Nice, France